CLINICAL TRIAL: NCT00475267
Title: An Observational, Prospective Evaluation of the Trifecta Valve
Brief Title: Aortic Valve Replacement With Trifecta(TM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0601
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Insufficiency; Regurgitation, Aortic Valve; Aortic Valve Incompetence; Aortic Valve Stenosis
Keywords: aortic valve; heart valve; tissue valve; bioprosthesis; valve disorder; valve disease; cardiac surgery; aortic valve stenosis; aortic valve regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Trifecta aortic heart valve — Intended as a replacement for a diseased, damaged, or malfunctioning aortic heart valve.

SUMMARY:
The purpose of this study is to confirm the clinical safety and effectiveness of the Trifecta valve.

DETAILED DESCRIPTION:
The clinical investigation is a multi-center, multi-country, prospective, non-randomized, observational study designed to evaluate the safety and effectiveness of the Trifecta valve.

ELIGIBILITY:
Inclusion Criteria:

* Requires aortic valve replacement (heart surgery such as bypass is allowed at the same time).
* Legal age.
* Signed informed consent prior to surgery.
* Willing to complete all follow-up requirements.

Exclusion Criteria:

* Pregnant or nursing women.
* Have already had a valve replaced other than the aortic valve.
* Needs another valve replaced.
* Cannot return for required follow-up visits.
* Have active endocarditis.
* Acute preoperative neurological event (such as a stroke).
* Renal dialysis.
* History of substance abuse within one year, or a prison inmate.
* Participating in another study.
* Life expectancy less than two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Characterize patient NYHA functional classification status. | At required follow-up intervals
Characterize the hemodynamic performance of the valve. | At required follow-up intervals
Establish adverse event rates. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Hartzell Schaff, MD, Principal Investigator — Mayo Clinic
Locations (5):
- Canada (5):
  - University of British Columbia, St. Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hôpital Laval, Québec, Quebec